CLINICAL TRIAL: NCT00959218
Title: Multi-centre, Randomized, Double-blind, Placebo-controlled Study to Investigate the Efficacy and Safety of the Pain Relieving Effect of Dronabinol in Patients With Multiple Sclerosis Associated With Central Neuropathic Pain
Brief Title: Efficacy and Safety of the Pain Relieving Effect of Dronabinol in Central Neuropathic Pain Related to Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bionorica Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: cnp-MS-0601 / MC-2006-01
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Central Neuropathic Pain in Multiple Sclerosis
Keywords: Dronabinol; (-)trans-delta9-tetrahydrocannabinol; central neuropathic pain; multiple sclerosis; analgesic; Central neuropathic pain related to multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dronabinol (Experimental)
  Interventions: Drug: Dronabinol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dronabinol — oral solution, daily dose up to 15 mg, treatment up to 2.5 years
  Other Names: (-)trans-delta9-tetrahydrocannabinol
  Arms: Dronabinol
Drug: Placebo — oral solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Dronabinol is effective and safe in relieving central neuropathic pain in multiple sclerosis patients.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is in all probability an autoimmune disease causing severe neurological disability due to inflammation and degeneration in the central nervous system (CNS). MS affects over 1 million people worldwide. Central neuropathic pain is associated with approximately 30% of all patients with MS. MS-accompanying pain has a major impact on the patients' quality of life as usual conventional analgesics are little effective. The aim of this clinical study is to determine whether Dronabinol is effective and safe in relieving central neuropathic pain in multiple sclerosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis acc. to McDonald diagnostic criteria
* EDSS score between 3 and 8 (incl.)
* Patients who are in a stable phase of multiple sclerosis
* Patients with MS-related central neuropathic pain for at least 3 months

Exclusion Criteria:

* Severe concomitant diseases
* Certain concomitant therapies (in particular: pain influencing concomitant therapies)
* Dronabinol intake within the last 12 months prior to study entry or Marihuana use within one month prior to study entry

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2007-06; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Mean change of baseline pain severity score on the 11-point Likert Numerical Rating Scale recorded in patient diary | max. 2.5 years

SECONDARY OUTCOMES:
Likert Numerical Rating Scale pain relief | max. 2.5 years
Pain-related sleep interference | max. 2.5 years
SF-36 (QoL-questionnaire) | max. 2.5 years
Intake of rescue medication | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Schimrigk, MD, Principal Investigator — Klinikum Luedenscheid
Locations (1):
- Maerkische Kliniken GmbH, Klinikum Luedenscheid, Akademisches Lehrkrankenhaus der Universitaet Bonn, Klinik fuer Neurologie, Lüdenscheid, Germany